CLINICAL TRIAL: NCT03021044
Title: Physical Activity Intervention for Patients With Reduced Physical Performance After Acute Coronary Syndrome: a Randomized Clinical Trial (The HULK Pilot Study).
Brief Title: Physical Activity Intervention for Patients With Reduced Physical Performance After Acute Coronary Syndrome
Acronym: HULK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Interventional cardiologist and Associate Professor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 161098
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STANDARD OF CARE (Other): The standard of care group will be recommended about medications and a correct life style (physical activity, low salt and low fat diet, no smoking) in order to prevent cardiovascular events. In this 15-minutes talk study doctor will explain to patients and relatives the importance of aerobic physical activity (30-60 minutes daily, moderate intensity, for example speedy walking, for at least 5 days/weekly) with the aim of reducing cardiovascular risk. Patients will also receive a brochure with clear explanations. Study doctor and study coordinator will be helpful for any question and they will ensure that patients and relatives understand the importance of physical activity for cardiovascular health.
  Interventions: Other: standard of care
- PHYSICAL ACTIVITY INTERVENTION (Experimental): Besides standard of care, the experimental group will participate to a program of physical activity intervention. Following hospital discharge, participants in stable clinical conditions will be referred by their cardiologist to the exercise-based secondary prevention program. All exercise testing and training sessions will be performed without discontinuing the prescribed medications. On admission to the program, and quarterly during follow-up, each patient will perform a 1-km treadmill walk test as previously described (1k-TWT).
  Interventions: Other: physical activity intervention

INTERVENTIONS:
Other: physical activity intervention — 30, 60, 90 and 120 days after hospital discharge a clinical visit and session of physical activity training and program
  Arms: PHYSICAL ACTIVITY INTERVENTION
Other: standard of care — 30, 60, 90 and 120 days after hospital discharge a clinical visit with correct style life recommendation
  Arms: STANDARD OF CARE

SUMMARY:
RATIONALE AND OBJECTIVE OF THE STUDY

Patients with low functional capacity (frail patients) with cardiovascular disease, in particular those undergoing invasive procedures or suffering from coronary artery disease, have a much higher adverse events, death and re-hospitalizations. and complications, suggesting the need for a more accurate functional stratification and a more careful evaluation of the risk/benefit ratio of some invasive procedures. An early and ad hoc physical activity intervention could be improve functional autonomy of these patients early after discharge with benefit on long-term outcome. The present study is performed to assess the impact, evaluated by Short Physical Performance Battery (SPPB), of a program of physical activity early after discharge in elderly patients aged 75 years and older with low physical performance.

This is an interventional, multicenter, prospective, randomized, phase III study. The present study is expected to enroll elderly patients admitted to hospital for acute coronary syndrome undergoing percutaneous coronary angioplasty and stratified with SPPB score predischarge. At the moment of discharge there will be a screening: patients with SPPB score 0-2 o 10-12 will be exclusively followed up by clinical visit every year. Patients with SPPB score 3-9 will be evaluated during the inclusion visit when SPPB will be repeated. If SPPB score will be 0-3 or 10-12, patients will be considered screening failure and will be followed up by clinical visit; patients with SPPB score between 4 to 9 will be randomized to standard of care (see below) or to an ad hoc physical activity program (see below). The aim of the study is to demonstrate 6 months later an improvement in the SPPB score (at least 1 point) in patients randomized to physical activity intervention versus patients randomized to standard of care. All patients will be evaluated until 3 years after randomization.

DETAILED DESCRIPTION:
BACKGROUND Physical activity helps to prevent stroke, type II diabetes mellitus and coronary artery disease, while physical inactivity has been linked to declines in both muscle strength and cardiovascular function. Despite the evidence of the benefits of physical activity are well known, 61% of adults over the age of 65 are not meeting the recommended levels of physical activity. It has been demonstrated that regular physical exercise benefits in primary and secondary prevention in patients with cardiovascular diseases and improves functional capacity. The incidence of cardiovascular disease is higher in older patients (especially over 75 years old). In Italy, life expectancy at birth has reached 80 years in men and 85 in women; in about 50 years, life expectancy at the age of 80 has increased by an extraordinary 61% and 55%, respectively, due to more effective therapies and lower mortality of many diseases. So, as recommended by guidelines, physical activity should be suggested to older coronary patients; some studies demonstrated the benefit of physical training also in older patients, but only few studies enrolled patients aged 65 years and over because of some difficulties about patients' compliance mainly due to logistic problems and lack of motivation by doctors. As far as we know no studies have evaluated impact of physical activity intervention on functional capacity of older patients admitted to hospital for acute coronary syndrome. Among the numerous tests proposed in the literature for the functional evaluation and objective measures of physical capability in elderly patient, the Short Physical Performance Battery (SPPB) and the evaluation of hand grip strength (grip strength) are those characterized by an improved prognostic ability and an easy administration.

RATIONALE AND OBJECTIVE OF THE STUDY Patients with low functional capacity (frail patients) with cardiovascular disease, in particular those undergoing invasive procedures or suffering from coronary artery disease, have a much higher adverse events, death and re-hospitalizations. and complications, suggesting the need for a more accurate functional stratification and a more careful evaluation of the risk/benefit ratio of some invasive procedures. An early and ad hoc physical activity intervention could be improve functional autonomy of these patients early after discharge with benefit on long-term outcome. The present study is performed to assess the impact, evaluated by Short Physical Performance Battery (SPPB), of a program of physical activity early after discharge in elderly patients aged 75 years and older with low physical performance.

STUDY DESIGN This is an interventional, multicenter, prospective, randomized, phase III study. The present study is expected to enroll elderly patients admitted to hospital for acute coronary syndrome undergoing percutaneous coronary angioplasty and stratified with SPPB score predischarge. At the moment of discharge there will be a screening: patients with SPPB score 0-2 o 10-12 will be exclusively followed up by clinical visit every year. Patients with SPPB score 3-9 will be evaluated during the inclusion visit when SPPB will be repeated. If SPPB score will be 0-3 or 10-12, patients will be considered screening failure and will be followed up by clinical visit; patients with SPPB score between 4 to 9 will be randomized to standard of care (see below) or to an ad hoc physical activity program (see below). The aim of the study is to demonstrate 6 months later an improvement in the SPPB score (at least 1 point) in patients randomized to physical activity intervention versus patients randomized to standard of care. All patients will be evaluated until 3 years after randomization.

RANDOMIZATION

At discharge an investigator doctor and a study coordinator show to patients the study protocol, aims, risks and benefit. If the patient accepts to participate to the study, he signs the informed consent and he will be evaluated with SPPB score and other tests in the screening evaluation (T0). Patients with SPPB score <3 or >9 will be excluded and will be followed up with exclusively clinical visit every year. Patients with SPPB score 4-9 will be enrolled and data will be collected in the study case report form. These patients will be re-evaluated in the inclusion visit 30 days later (T1); if SPPB score will be 0-3 or 10-12 the patients will be considered screening failure and they will be followed up exclusively with clinical visit every year; on the contrary, if SPPB score will be 4-9, patients will be randomized to standard of care group or experimental group. There will be a stratified randomization by:

* male vs. female
* SPPB value 4-6 vs. SPPB value 7-9
* admission for ST-segment elevation myocardial infarction vs. non ST-segment elevation acute coronary syndrome

DESCRIPTION OF THE STUDY GROUPS

* STANDARD OF CARE GROUP The standard of care group will be recommended about medications and a correct life style (physical activity, low salt and low fat diet, no smoking) in order to prevent cardiovascular events. In this 15-minutes talk study doctor will explain to patients and relatives the importance of aerobic physical activity (30-60 minutes daily, moderate intensity, for example speedy walking, for at least 5 days/weekly) with the aim of reducing cardiovascular risk. Patients will also receive a brochure with clear explanations. Study doctor and study coordinator will be helpful for any question and they will ensure that patients and relatives understand the importance of physical activity for cardiovascular health.
* EXPERIMENTAL GROUP, PHYSICAL ACTIVITY INTERVENTION Besides standard of care, the experimental group will participate to a program of physical activity intervention. Following hospital discharge, participants in stable clinical conditions will be referred by their cardiologist to the exercise-based secondary prevention program in dedicated centers. All patients should report no difficulty climbing one flight of stairs without resting or performing basic activities of daily living. The ultimate goal of the program is long-term promotion and maintenance of a physically active lifestyle in order to improve cardiorespiratory fitness and functional ability. Patients will be treated for cardiovascular and other diseases according to accepted international guidelines. All exercise testing and training sessions will be performed without discontinuing the prescribed medications. On admission to the program, and quarterly during follow-up, each patient will perform a 1-km treadmill walk test as previously described. Briefly, the test will be carried out as follows: the participants will be instructed to select a pace that they could maintain for 10 to 30 min at a moderate perceived exercise intensity using the Borg 6-20 scale. Participants will start the test walking on the level at 2.0 km/h, with subsequent increases of 0.3 km/h every 30 s up to a walking speed corresponding to a perceived exertion of 11-13 on the Borg scale. The test will be then started and the rate of perceived exertion acquired every 2 min. Walking speed will be adjusted to maintain the selected moderate perceived intensity. Heart rate will be monitored continuously during the test. Blood pressure will be monitored at least before and immediately after the test. No individual will be excluded on the basis of his/her performance on the treadmill protocol. Subjects walking at a perceived moderate speed < 3.0 km/h will perform the test over the distance of 500-m. The time to complete either 500-m and 1-km will be recorded and averaged walking speed calculated accordingly.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age ≥70 years old
* hospital admission for acute coronary syndrome
* coronary artery angiography and successfully percutaneous coronary revascularization
* result of the short physical performance battery test at the inclusion visit between 4 and 9

Exclusion Criteria:

* chronic heart failure (new york heart association classification III-IV)
* left ventricle ejection fraction <30%.
* severe aortic or mitral valvulopathy
* three vessel coronary artery disease or left main coronary artery disease requiring surgical coronary revascularization
* need of staged percutaneous coronary intervention
* severe cognitive impairment (defined as short portable mental status questionnaire < 4)
* physical limitation/impairment not permitting physical activity training annd program
* life expectancy <12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Physical performance | 6 months
  result of the short physical performance battery test

SECONDARY OUTCOMES:
Physical performance | 1 year
  result of the short physical performance battery test
Physical performance | 2 years
  result of the short physical performance battery test
Physical performance | 3 years
  result of the short physical performance battery test
clinical adverse events | 1 year
  cumulative occurrence of all-cause mortality and all-cause hospital readmission
clinical adverse events | 2 years
  cumulative occurrence of all-cause mortality and all-cause hospital readmission
clinical adverse events | 3 years
  cumulative occurrence of all-cause mortality and all-cause hospital readmission
cardiac adverse events | 1 year
  cumulative occurrence of cardiovascular death and hospital readmission for cardiovascular cause
cardiac adverse events | 2 years
  cumulative occurrence of cardiovascular death and hospital readmission for cardiovascular cause
cardiac adverse events | 3 years
  cumulative occurrence of cardiovascular death and hospital readmission for cardiovascular cause

OTHER OUTCOMES:
compliance to antiplatelet agents | 1 year
  percentage of patients maintaining dual antiplatelet regimen
physical training and session side effects | 6 months
  cumulative occurrence of any complications or adverse events during the physical activity training and session

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - University Hospital of Ferrara, Cona, Ferrara
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Ospedale Santa maria delle Croci, Ravenna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raisi A, Zerbini V, Myers J, Piva T, Campo G, Mazzoni G, Grazzi G, Mandini S. A Novel Motivational Approach in the Management of Older Patients With Cardiovascular Disease. J Cardiopulm Rehabil Prev. 2023 Jul 1;43(4):309-310. doi: 10.1097/HCR.0000000000000791. Epub 2023 Apr 5. No abstract available. PMID 37014940
- [Derived] Erriquez A, Pavasini R, Biscaglia S, Tebaldi M, Tonet E, Maietti E, Cimaglia P, Grazzi G, Scoccia A, Cardelli LS, Verardi FM, Morelli C, Campana R, Rubboli A, Mazzoni G, Volpato S, Ferrari R, Campo G. The impact of periprocedural myocardial infarction on mortality in older adults with non-ST-segment elevation acute coronary syndrome: a pooled analysis of the FRASER and HULK studies. J Cardiovasc Med (Hagerstown). 2021 Jul 1;22(7):546-552. doi: 10.2459/JCM.0000000000001146. PMID 34076602
- [Derived] Campo G, Tonet E, Chiaranda G, Sella G, Maietti E, Bugani G, Vitali F, Serenelli M, Mazzoni G, Ruggiero R, Villani G, Biscaglia S, Pavasini R, Rubboli A, Campana R, Caglioni S, Volpato S, Myers J, Grazzi G. Exercise intervention improves quality of life in older adults after myocardial infarction: randomised clinical trial. Heart. 2020 Nov;106(21):1658-1664. doi: 10.1136/heartjnl-2019-316349. Epub 2020 Mar 6. PMID 32144189
- [Derived] Tonet E, Maietti E, Chiaranda G, Vitali F, Serenelli M, Bugani G, Mazzoni G, Ruggiero R, Myers J, Villani GQ, Corvi U, Pasanisi G, Biscaglia S, Pavasini R, Lucchi GR, Sella G, Ferrari R, Volpato S, Campo G, Grazzi G. Physical activity intervention for elderly patients with reduced physical performance after acute coronary syndrome (HULK study): rationale and design of a randomized clinical trial. BMC Cardiovasc Disord. 2018 May 21;18(1):98. doi: 10.1186/s12872-018-0839-8. PMID 29783928